CLINICAL TRIAL: NCT04745468
Title: Selective Depletion of C-reactive Protein by Therapeutic Apheresis (CRP Apheresis) After Elective Primary Coronary Bypass Surgery
Brief Title: Study on CRP Apheresis After Coronary Bypass Surgery
Acronym: CABY1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentracor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02 CABY1
Record Dates: First submitted 2020-12-03; First posted 2021-02-09 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-02

CONDITIONS: Post-cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apheresis Group (Experimental): 20 patients receive 2 apheresis treatments at intervals of 24 ± 12 h (additionally to the standard therapy after bypass surgery). The first treatment starts within 24 h postoperatively. If the CRP concentration increases to at least 30 mg/L 6-18 h after the end of the second treatment, a third treatment is performed.
  For each treatment the 1 - 2.5-fold plasma void is processed. The duration of each treatment is 4-6 h.
  Interventions: Device: CRP apheresis
- Control group (No Intervention): 17 patients of the control group receive the standard therapy after bypass surgery.

INTERVENTIONS:
Device: CRP apheresis — Selective CRP apheresis by use of the PentraSorb-CRP adsorber
  Arms: Apheresis Group

SUMMARY:
The CABY1 study is conducted open, controlled, randomized and monocentric. The efficacy and tolerability of CRP apheresis in patients undergoing elective primary coronary bypass surgery is investigated.

DETAILED DESCRIPTION:
CABY1 is a clinical trial to study the reduction of C-reactive protein (CRP) by therapeutic apheresis (CRP apheresis) in patients undergoing elective primary coronary bypass surgery.

The term therapeutic apheresis describes therapeutical procedures whose effect is based on the elimination of blood components with a pathogenic function within the disease process. Elimination takes place in adsorbers outside the body in an extracorporeal circuit. To remove the pathogenic substances, blood plasma is separated from the circuit and passed through an adsorber. The purified blood plasma is then reunited with the solid blood components and returned to the patient.

The "PentraSorb® CRP" adsorber used for CRP apheresis is CE-certified. It serves for the selective depletion of the C-reactive protein from human plasma.

As a cause of the damaging effect of the C-reactive protein it is assumed that the CRP as an inflammatory mediator favours the destruction of cardiac muscle tissue (in conjunction with complement) and has a negative influence on the regeneration of the traumatized tissue.

The aim of the CABY1 study is to investigate if the tissue damage of the heart can be reduced by depletion of the C-reactive protein after elective coronary bypass surgery. A possible protective effect of CRP apheresis will be determined from laboratory biomarkers (e.g., troponin I, CM-MB, IL-6) and cardiac events.

20 randomly selected patients receive apheresis treatments with a duration of 4-6 h each the following 2-3 days after bypass surgery, the 20 patients of the controls do not receive apheresis. The biomarkers required for the evaluation of the treatment success are determined over a period of 4 days after surgery on the basis of the routine blood tests. Cardiac events are documented until the patient is discharged.

ELIGIBILITY:
Inclusion Criteria:

* elective, isolated, primary coronary bypass surgery
* 2 or 3-fold CHD with or without main stem stenosis
* Obtained LVEF (> 30%, trans-oesophageal echocardiography (TEE) or angiography)
* Heart-lung machine (HLM; 'two-stage' cannulation)
* Antegrade Bretschneider cardioplegia
* Mild hypothermia (32 °C)
* Standard anesthesia (isoflurane)
* Intraoperative standard protocol (500 mg ASA after 2 h, low dose heparinization after 4 h)
* written informed consent
* legal capacity

Exclusion Criteria:

Preoperatively

* PCI (within last 2 weeks)
* Renal insufficiency (creatinine > 1.3 mmol/L or requiring dialysis)
* Combination interventions
* Re-surgery
* Emergency of urgent surgery indication
* Acute coronary syndrome (IAP, NSTEMI, STEMI)
* Preoperatively positive hs-troponin I > 40 ng/ml
* Chronic arterial fibrillation
* Acute infectious disease (body temperature > 38.0°C)
* Systolic blood pressure < 100 mmHg
* Known hypersensitivity to therapeutic apheresis
* Cardiac shock
* Pregnancy or lactation
* Participation in other interventional trial

During surgery

* Radialis removal
* Coronary TEA (if blood flow within bypass < 20 ml/min)
* Off-pump
* Hemofiltration
* Combination intervention (e.g. mitral valve reconstruction, LAA)
* Maze procedure
* Bypass low-flow closure, ECG changes
* Antithrombotic therapy (intraoperative clopidogrel and/or aspirin)
* Second HLM
* Second cardioplegic cardiac arrest
* Intraaortal balloon pumping / balloon pulsation (IABP)
* Extracorporeal membrane oxygenation (ECMO)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Tissue damage of the heart | Every 24 hours for up to 96 hours after bypass surgery
  Daily determination of the concentration of the biomarker Troponin I (hsTnI)

SECONDARY OUTCOMES:
Safety of CRP apheresis | 24 hours after each apheresis
  Incidence of expected and unexpected adverse effects
Cardiac events | Until the patient is discharged from the hospital, an average of 7 days
  Documentation of cardiac events:
  * Cardiac arrythmias
  * Perioperative myocardial infarction (PMI)
  * Cardiopulmonary resuscitation (CPR)
  * Low cardiac output syndrome (LCOS)
  * Re-surgery
  * Percutaneous coronary intervention (PCI)
  * Angina pectoris
Tissue damage of the heart with Procalcitonin | Every 24 hours for 72 hours after bypass surgery
  Daily determination of the concentration of:
  - Procalcitonin
Tissue damage of the heart with CK-MB | Every 24 hours for 72 hours after bypass surgery
  Daily determination of the concentration of:
  - Creatine kinase, MB fraction (CK-MB)
Tissue damage of the heart with Myoglobin | Every 24 hours for 72 hours after bypass surgery
  Daily determination of the concentration of:
  - Myoglobin
Tissue damage of the heart with Leukocytes | Every 24 hours for 72 hours after bypass surgery
  Daily determination of the concentration of:
  - Leukocytes
Tissue damage of the heart with Interleukin-6 | Every 24 hours for 72 hours after bypass surgery
  Daily determination of the concentration of:
  - Interleukin-6 (IL-6)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Thielmann, Prof. Dr. med., Principal Investigator — Westdeutsches Herz- und Gefäßzentrum Essen, Klinik für Thorax- und Kardiovaskuläre Chirurgie
Locations (1):
- Klinik für Thorax- und Kardiovaskuläre Chirurgie, Essen, Germany

IPD SHARING:
Plan to Share IPD: No